CLINICAL TRIAL: NCT05796531
Title: Therapeutic Evaluative Conditioning to Reduce Adolescents' Self-injurious Thoughts and Behaviors During and After Psychiatric Inpatient Hospitalization
Acronym: TEC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Franciscan Hospital For Children, INC. (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Harvard University (Other)
Responsible Party: Principal Investigator, Kelly Zuromski, Director of Research, Franciscan Hospital For Children, INC.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R34MH124973-01 (NIH)
Record Dates: First submitted 2023-02-06; First posted 2023-04-03 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Self-Injurious Behavior; Suicidal Ideation; Suicide Attempts
MeSH Terms: conditions — Self-Injurious Behavior; Suicidal Ideation; Suicide, Attempted

STUDY DESIGN:
Intervention Model Description: Intervention and control arms
Who Masked: Participant
Masking Description: Participants will not know which group they are in but researchers will know.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active intervention arm (Active Comparator): Participants will complete the intervention on a mobile device.
  Interventions: Behavioral: Therapeutic Evaluative Conditioning
- Control arm (Sham Comparator): Participants will complete the sham comparator on a mobile device.
  Interventions: Behavioral: Neutral comparison condition

INTERVENTIONS:
Behavioral: Therapeutic Evaluative Conditioning — Participants are told which pictures are "matched pairs." They find the "matched pairs" among 4 or 8 pictures. By associating pictures and words associated with SITB (e.g., pictures of cut skin, pictures of people engaging in potentially suicidal behaviors, and the word "death") with naturally aversive images (e.g., snakes and spiders), it increases the aversion to SITB. The second goal is to increase liking toward the self by pairing self-relevant stimuli (e.g., the participant's name or other self-relevant details, as well as words like "I" and "me").
  Arms: Active intervention arm
Behavioral: Neutral comparison condition — Match neutral pictures to account for doing an intervention.
  Arms: Control arm

SUMMARY:
Suicide is the 2nd leading cause of death among adolescents, with the highest risk period for suicide being the month following psychiatric inpatient hospitalization. The investigators propose testing a brief, scalable intervention using evaluative conditioning aimed at reducing suicidal thoughts and behaviors among adolescents during and after inpatient hospitalization. Scalable interventions, such as the one proposed that reduce suicide risk during this markedly high-risk period, could result in large-scale decreases in suicide death.

DETAILED DESCRIPTION:
The project has two phases: a pilot phase and randomized controlled trial phase. The study within each phase consists of three parts: an inpatient study period, where baseline data are collected, the intervention is initiated, and treatment targets and outcomes are assessed; a one-month post-discharge period, where the intervention is continued and treatment targets and outcomes are assessed and a one-month post-intervention period, where the intervention is no longer administered but treatment targets and outcomes are assessed to test whether the intervention has sustained treatment effects. For the inpatient period, the intervention and the assessment of the treatment targets and outcomes will each be delivered via an iPad administered by a research assistant (RA). During the post-discharge and post-intervention periods assessments will be administered via smartphone mobile apps.

A. Inpatient period. There are eight components to the inpatient part of the study: (1) Parent informed consent and permission. As close as possible to the patient's intake, parents will provide consent and permission for their child to participate. For patients over the age of 17, the patient will be able to provide consent for themselves. For all participants, the investigators will obtain parent consent to collect the qualitative data from the parent on their child's experience of the intervention. (2) Patient assent and baseline data collection. As part of standard clinical intake on the McLean-Franciscan inpatient unit, participants will complete a self-report version of the Self-Injurious Thoughts and Behaviors Interview (SITBI), which will be integrated into the study data set. As soon as possible following parental consent, study staff will meet with participant to obtain assent and collect baseline data. Patient baseline data collection will consist of administration of study measures, including explicit and implicit measures of aversion toward SITB-related and self-related stimuli (i.e., baseline assessments of the treatment target), SITB since admission will be assessed (assuming it is more than 1 day after completing the full SITBI) using a "since last assessment" version of the SITBI, and a brief interview to gather information that can will be used to personalize the TEC intervention, such as details regarding methods the patient has thought of or used to self-injure. Researchers will also schedule a time for patients to complete TEC each day of their inpatient stay. (3) Personalize TEC. Following, the interview, for participants' in the active TEC arm, researchers will setup TEC to be personalized for each participant. For example, the investigators will enter the participants' name in the positive-self TEC intervention based on studies showing that evaluative conditioning paradigms where first names are paired with positive stimuli have been shown to improve implicit affect to self-related stimuli. (4) Installation of apps on patient's phone for the post-discharge part of the study. Parents bring the patient's smartphone to the hospital. The investigators have developed procedures to facilitate receiving and returning patients' phones, such as texting parents reminders and having lockboxes available for phone drop-off and pickup. An app will be installed on participants' phone. (5) TEC intervention and pre/post ratings relevant to acceptability. Because electronic devices, such as phones or tablets, are not allowed on the inpatient unit, each day a RA will bring an iPad to the patient to complete (a) the TEC intervention and (b) pre-/post-intervention measurements of mood, desire to die and urge to kill oneself to help evaluate the acceptability of TEC. (6) Assessment of treatment target and burdensomeness of the intervention. Every three days on the inpatient unit, participants will also complete measures of explicit and implicit aversion to SITB- and self-related stimuli, which are the treatment targets and ratings of the burdensomeness of TEC to evaluate the feasibility of TEC. (7) Assessment of the outcome. Daily, prior to completing the TEC intervention, participants will complete a questionnaire regarding the occurrence of any SITB in the prior 24 hours. SITBs are assessed frequently for the purposes of accurate measurement, such that participants do not have to be remember SITB events over a few days. Daily sessions will take less than 10 minutes. (8) Qualitative interview of intervention experiences. Every three days, a brief interview will assess participants' experiences and reactions to the intervention and qualitatively assess their mood and suicidal thoughts.

B. Post-discharge intervention period. For 28 days after discharge, participants will receive daily push notifications to complete a brief survey regarding SITB in the past 24 hours, the TEC intervention, and pre-/post-intervention mood, desire to die and urge to kill oneself. The push notification will be sent in the morning; additional reminders will be sent throughout the day until the tasks are completed with a maximum of 5 reminders. Once every two weeks, participants will also be asked to complete (1) implicit cognition measures to assess the treatment target and (2) a brief measure regarding the burdensomeness of TEC. A RA will contact the participant after two consecutive days of non-compliance.

C. Post-intervention follow-up. Two- and four-weeks after TEC has ended, the investigators will assess implicit cognitions (i.e., the treatment target) and SITB to test whether treatment effects persist without the intervention. The investigators will send reminders and contact participants if they do not complete the assessments.

ELIGIBILITY:
Inclusion Criteria:

* Be a patient on McLean-Franciscan Child and Adolescent Inpatient Program (MF-CAIP) of Franciscan Children's (FC)
* Be 12-19 years-old
* Own a smartphone
* Have a parent/guardian that can provide permission
* Child can assent
* Presentation to the hospital with non-suicidal self-injury (NSSI), suicidal ideation or a suicide attempt.

Exclusion Criteria:

* Any factor that impairs an individual's ability to comprehend and effectively participate in the study, including
* an inability to speak or write English fluently
* the presence of gross cognitive impairment due to florid psychosis, intellectual disability, dementia, acute intoxication, etc., or the presence of extremely agitated or violent behavior
* a potential discharge location anticipated to be a residential program in which the average length of stay is more than 14 days

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 155 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Self-injurious thoughts and behaviors | During inpatient hospitalization (average 14 days), plus an additional two months post- hospitalization.
  The investigators will assess the presence and frequency of non-suicidal self-injury, suicidal thoughts, suicide plans, suicide attempts and other suicidal behaviors, such as aborted suicide attempts. The investigators will also assess the severity of suicidal thoughts as well.

CONTACTS AND LOCATIONS:
Locations (1):
- Franciscan Hospital For Children, Inc., Brighton, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the guidelines of this funding opportunity announcement (FOA), all data will be shared via the National Database for Clinical Trials related to Mental Illness (NDCT) and the National Institute of Mental Health Data Archive (NDA).
  Raw (descriptive) data. The investigators will share all baseline data, summaries from behavioral tasks (i.e., Affect Misattribution Procedure) and intervention (Therapeutic Evaluative Conditioning), follow-up data, and real-time monitoring data. These data will be linked by Globally Unique Identifier (GUID) and stored in comma separated variable (CSV) format. A formal "data expected list" will be created within six months of award, as required by the FOA.
Supporting Information: Analytic Code
Time Frame: Twice yearly.
Access Criteria: public
URL: https://nda.nih.gov/

REFERENCES:
- [Background] Franklin JC, Fox KR, Franklin CR, Kleiman EM, Ribeiro JD, Jaroszewski AC, Hooley JM, Nock MK. A brief mobile app reduces nonsuicidal and suicidal self-injury: Evidence from three randomized controlled trials. J Consult Clin Psychol. 2016 Jun;84(6):544-57. doi: 10.1037/ccp0000093. Epub 2016 Mar 28. PMID 27018530